CLINICAL TRIAL: NCT02984306
Title: Effect of Cherry Powder Supplementation on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 115229/01
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary supplement (Experimental)
  Interventions: Dietary Supplement: Cherry powder; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cherry powder
Dietary Supplement: Placebo

SUMMARY:
Examining the effect of four weeks of cherry powder supplementation on flow mediated dilatation

ELIGIBILITY:
Inclusion Criteria:

* physically inactive no prescription medications

Exclusion Criteria:

* physically active taking prescription medication

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation | change from baseline to 4 weeks dietary supplementation

SECONDARY OUTCOMES:
Plasma nitrite concentration | change from baseline to 4 weeks dietary supplementation
Plasma nitrate concentration | change from baseline to 4 weeks dietary supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Sport & Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No